CLINICAL TRIAL: NCT04230954
Title: A Phase II Study of Cabozantinib (XL184) Plus Pembrolizumab for Recurrent, Persistent and/or Metastatic Cervical Cancer
Brief Title: Cabozantinib Plus Pembrolizumab for Recurrent, Persistent and/or Metastatic Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of South Alabama (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-67-MCI-1001
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Cervical Cancer; Recurrent Cervical Cancer; Metastatic Cervical Cancer; Persistent Cervical Cancer
Keywords: Recurrent Cervical Cancer; Cervical Cancer; Cervical Carcinoma; PD L1 positivity; Immunotherapy; Squamous Carcinoma; Adenocarcinoma; Adenosquamous Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Adenosquamous | interventions — cabozantinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (XL 184) Plus Pembrolizumab (Experimental): A Phase II Study of Cabozantinib (XL 184)Plus Pembrolizumab for Recurrent, Persistent and/or Metastatic Cervical Cancer
  Interventions: Drug: Cabozantinib 40 MG oral once a day; Drug: Pembrolizumab 200 mg IV every 3 weeks

INTERVENTIONS:
Drug: Cabozantinib 40 MG oral once a day — Cabozantinib 40 mg oral once a day
  Other Names: Cabometyx
Drug: Pembrolizumab 200 mg IV every 3 weeks — Pembrolizumab 200 mg IV every 3 weeks
  Other Names: Keytruda

SUMMARY:
Drug: Cabozantinib Drug: Pembrolizumab

DETAILED DESCRIPTION:
This study is a multi-center, single arm, open label trial to evaluate the efficacy and safety of Cabozantinib (XL184) plus Pembrolizumab in recurrent, persistent and/or metastatic cervical cancer with PD-L1 tumor positivity.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent cervical cancer after prior systemic chemotherapy for which there is no curative intent option
* Documented histologic cervical cancer (acceptable histologies: squamous carcinoma, adenocarcinoma, and adenosquamous carcinoma)
* Patients must have PD-L1 tumor positivity as defined as CPS>/= 1
* Age greater than 18 and ECOG performance status of <= 2
* Adequate organ and marrow function

Exclusion Criteria:

* Prior treatment with cabozantinib or pembrolizumab
* Receipt of any type of small molecule kinase inhibitor
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery
* Anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel)
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions: Cardiovascular disorders: Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias Uncontrolled hypertension despite optimal antihypertensive treatment, stroke
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose
* Active autoimmune disease requiring systemic therapy within the past 2 years
* Active infection requiring systemic therapy within the past month
* History of immunodeficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 24 months
  Six months progression free survival as defined by RECIST v1.1 measured from signed written consent to the date of first documented tumor progression using RECIST v1.1, or death due to any cause or 24 months after the end of study treatment.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 24 months
  Overall response defined by Response Evaluation Criteria in Solid Tumors (RECIST v.1.1 criteria).
Overall Survival | Up to 24 months
  Overall survival will be defined as the time from signed written consent to the date of death or 24 months after the end of study treatment. A patient who has not died will be censored at the last known date of contact
Incidence of Emergent Adverse Events | Up to 6 Months
  Evaluate the safety and tolerability measured by incidence of adverse events and serious adverse events, deaths, and laboratory abnormalities as measured by Common Terminology Criteria for Adverse Events v.4.0
Cervical Cancer Quality of Life | Up to 6 Months
  Quality of life as assessed by FACT Cx quality of life questionnaire. This frequency questionnaire is scaled from 0-4 with 0 being not at all and 4 being very much.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie White, Study Director — University of South Alabama
Locations (1):
- University of South Alabama Mitchell Cancer Institute, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karim R, Jordanova ES, Piersma SJ, Kenter GG, Chen L, Boer JM, Melief CJ, van der Burg SH. Tumor-expressed B7-H1 and B7-DC in relation to PD-1+ T-cell infiltration and survival of patients with cervical carcinoma. Clin Cancer Res. 2009 Oct 15;15(20):6341-7. doi: 10.1158/1078-0432.CCR-09-1652. Epub 2009 Oct 13. PMID 19825956
- [Background] Yang W, Song Y, Lu YL, Sun JZ, Wang HW. Increased expression of programmed death (PD)-1 and its ligand PD-L1 correlates with impaired cell-mediated immunity in high-risk human papillomavirus-related cervical intraepithelial neoplasia. Immunology. 2013 Aug;139(4):513-22. doi: 10.1111/imm.12101. PMID 23521696
- [Background] Yakes FM, Chen J, Tan J, Yamaguchi K, Shi Y, Yu P, Qian F, Chu F, Bentzien F, Cancilla B, Orf J, You A, Laird AD, Engst S, Lee L, Lesch J, Chou YC, Joly AH. Cabozantinib (XL184), a novel MET and VEGFR2 inhibitor, simultaneously suppresses metastasis, angiogenesis, and tumor growth. Mol Cancer Ther. 2011 Dec;10(12):2298-308. doi: 10.1158/1535-7163.MCT-11-0264. Epub 2011 Sep 16. PMID 21926191
- [Background] Chung HC, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, Manzuk L, Piha-Paul SA, Xu L, Zeigenfuss S, Pruitt SK, Leary A. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Cervical Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2019 Jun 10;37(17):1470-1478. doi: 10.1200/JCO.18.01265. Epub 2019 Apr 3. PMID 30943124